CLINICAL TRIAL: NCT05455944
Title: Analgesic Efficacy of Pre-operative Oral Pregabalin in Dacryocystorhinostomy Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sameh Fathy (Other)
Responsible Party: Sponsor-Investigator, Sameh Fathy, Lecturer of anesthesia, ICU & pain management - Faculty of Medicine, Mansoura University
Organization: Mansoura University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Pregabalin in DCR surgery
Record Dates: First submitted 2022-07-10; First posted 2022-07-13 (Actual); Last update posted 2022-07-14 (Actual); Status verified 2022-07

CONDITIONS: Dacryocystitis
Keywords: Pregabalin; Dacryocystorhinostomy; Analgesia
MeSH Terms: conditions — Dacryocystitis; Agnosia | interventions — Pregabalin

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pregabalin Group (Active Comparator): Patients received two capsules: one at the night of surgery, and the other at 2 hours before the surgery
  Interventions: Drug: Pregabalin 150mg
- Control Group (Placebo Comparator): Patients received two capsules: one at the night of surgery, and the other at 2 hours before the surgery
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Pregabalin 150mg — Two capsules of pregabalin is administered orally to patients
  Other Names: Lyrica
  Arms: Pregabalin Group
Drug: Placebo — Two identical placebo capsules is administered orally to patients
  Other Names: Control
  Arms: Control Group

SUMMARY:
This study is conducted to evaluate the effects of preoperative oral pregabalin on postoperative pain and analgesic requirements in patients undergoing DCR surgery. The primary outcome is to compare pain scores by visual analogue scale (VAS). Secondary outcomes are the time of first analgesic request, the total analgesic requirements during the postoperative 24 hours, the incidence of PONV, in addition to effect on hemodynamic parameters between the two groups.

DETAILED DESCRIPTION:
External dacryocystorhinostomy (DCR) is still considered the golden standard for lacrimal surgery. It is a bypass technique which creates an anastomosis between the lacrimal sac and the nasal mucosa through a bony ostium via an external skin incision. External DCR can be completed under either local or general anesthesia. It is a painful surgical procedure that involves intra- and extra-ocular dissection, with a high prevalence post-operative nausea and vomiting (PONV). So, it is necessary to ensure a stress-free peri-operative period with adequate pain relief and a low incidence of PONV after DCR surgery.

Pregabalin is a lipophilic gamma-amino-butyric acid (GABA) analogue that binds to the voltage-gated calcium channels. It reduces the excitability of the dorsal horn neurons after tissue damage. It has anticonvulsant, anxiolytic and sleep-modulating properties. It was shown to be effective in several models of neuropathic pain, incisional injury, and inflammatory injury.

Preoperative administration of pregabalin is supposed to be a promising technique of enhancing postoperative pain control and reduction in postoperative opioid consumption.

This study is a prospective randomized double-blind clinical trial included 100 ASA I and II patients of both sex with age between 18 and 65 years old, who are planned for elective DCR surgery under general anesthesia in Mansoura University ophthalmology center. Informed written consent is obtained from all subjects in the study after ensuring confidentiality. Details of the anesthetic technique and the study protocol are clarified to the entire involved cases. Patients are randomly assigned to two equal groups according to computer-generated randomization schedule.

A prospective analysis of the collected data is performed using the Statistical Package for the Social Sciences (SPSS) program for Windows (version 22). All data are considered statistically significant if P value is ≤ 0.05.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiology (ASA) I and II patients.
* Scheduled for DCR surgery.

Exclusion Criteria:

* Patient' refusal of consent.
* Mental, psychological or neurological disorders.
* Patients with history of drug or alcohol abuse.
* History of know sensitivity to the used drugs.
* Bleeding or coagulation diathesis.
* Obese patients (body mass index (BMI) < 35).
* Pregnancy and lactation.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2020-12-30 (Actual); Study Completion 2021-12-30 (Actual)

PRIMARY OUTCOMES:
Changes in pain scores by visual analogue scale (VAS) | Up to 24 hours after the procedure
  Pain (VAS) score from 0 to 10 (0 = no pain and 10 = the worst imaginable pain)

SECONDARY OUTCOMES:
Changes in heart rate | Up to the end of the surgery
  Heart rate (beat/min) is recorded at five-minute intervals until the end of the surgery
Changes in mean arterial blood pressure | Up to the end of the surgery
  Blood pressure (mmHg) is recorded at five-minute intervals until the end of the surgery
First analgesic request | Up to 24 hours after the procedure
  The time of the first analgesic request for pethidine is recorded.
Total analgesic requirements of pethidine | Up to 24 hours after the procedure
  The amount of pethidine consumption given as a rescue analgesia to patients is measured all over the 24 hours.
Incidence of postoperative nausea and vomiting | Up to 24 hours after the procedure
  Incidence of postoperative nausea and vomiting is assessed up to 24 hours after the procedure

CONTACTS AND LOCATIONS:
Overall Officials: Sameh M Elsherbiny, MD, Study Director — Mansoura Faculty of Medicine
Locations (1):
- Department of Anesthesia, Mansoura University Hospitals, Al Mansurah, Dakahlia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No